CLINICAL TRIAL: NCT03168711
Title: Safety of Urate Elevation in Amyotrophic Lateral Sclerosis (ALS)
Acronym: SURE-ALS2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: The Salah Foundation (Other); Sean M. Healey & AMG Center for ALS (Other)
Responsible Party: Principal Investigator, Sabrina Paganoni, M.D., Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SURE-ALS2
Record Dates: First submitted 2017-05-24; First posted 2017-05-30 (Actual); Results first posted 2021-02-18 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS; Inosine; Uric acid; Urate; Glutathione; Biomarker; Oxidative stress; Oxidative damage
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Inosine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Inosine (Experimental): Subjects will be administered oral inosine daily. The dose of inosine will be titrated to obtain serum urate levels of 7 - 8 mg/dL.
  Interventions: Drug: Inosine
- Placebo (Placebo Comparator): Subjects will be administered oral placebo daily. The dose of placebo will be titrated to obtain serum urate levels of 7 - 8 mg/dL.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Inosine — Subjects on inosine will receive 1-6 capsules a day of 500 mg inosine titrated to target urate levels of 7 - 8 mg/dL.
  Arms: Inosine
Drug: Placebo — Subjects on placebo will receive 1-6 capsules a day of 500 mg placebo (sugar pill) titrated to target urate levels of 7 - 8 mg/dL.
  Arms: Placebo

SUMMARY:
This is a multi-center, 20-week study of inosine treatment.

Study Objectives and Endpoints The primary objective of the study is to determine the safety and tolerability of oral administration of inosine (administered daily) dosed to moderately elevate serum urate over 20 weeks.

The primary outcome measures will be

1. Safety, as measured by adverse events
2. Tolerability, defined as the ability of subjects to complete the entire 20-week study.

As an exploratory objective, we will test the feasibility and utility of a smartphone application for monitoring symptoms and disease progression in patients with amyotrophic lateral sclerosis (ALS).

DETAILED DESCRIPTION:
Amyotrophic lateral sclerosis (ALS) is a fatal, neurodegenerative disease for which there is no cure. Multiple lines of evidence have implicated oxidative stress in the pathophysiology of ALS. Urate (uric acid) is an endogenous antioxidant system, and urate may serve as a major defense against oxidative stress. Urate has emerged as a promising neuro-protectant and therapeutic target based on convergent epidemiological, laboratory, and clinical data in multiple neurodegenerative diseases, most notably Parkinson's disease (PD). In PD, urate elevation has been pursued as a potential therapy by administration of inosine, a urate precursor that is available as an over-the-counter supplement. Administration of inosine results in a predictable elevation of urate levels and has been shown to be safe and well tolerated in PD.

Analysis of ALS databases revealed that higher urate levels are an independent predictor of slower progression and prolonged survival in ALS. However, whether elevating urate in people with ALS would result in better outcomes is unknown.

The Principal Investigator has recently concluded a Pilot Study of Inosine in ALS, which was a short, open label, single center study involving 25 subjects [NCT02288091]. The study assessed safety and feasibility of urate elevation in patients with ALS. The Principal Investigator is now pursuing a multi-center Phase II trial to assess the findings of the open label study with longer exposure time.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-85.
2. Sporadic or familial ALS diagnosed as possible, laboratory-supported probable, probable, or definite as defined by revised El Escorial criteria (Appendix 1).
3. Slow vital capacity (SVC) ≥ 60% of predicted for age, height, and gender at the Screening Visit.
4. Capable of providing informed consent and following trial procedures.
5. Serum urate < 5.5 mg/dL at screening (i.e. below the population median serum urate levels).
6. Women must not be able to become pregnant (e.g. post menopausal, surgically sterile, or using adequate birth control methods) for the duration of the study and 3 months after study completion. Adequate contraception includes: abstinence, hormonal contraception (oral contraception, implanted contraception, injected contraception or other hormonal (patch or contraceptive ring, for example) contraception), intrauterine device (IUD) in place for ≥ 3 months, barrier method in conjunction with spermicide, or another adequate method.
7. Is able and willing to participate in the Mobile app study procedures.

Exclusion Criteria:

1. History of urolithiasis.
2. Urine pH < 5.5 at screening (as acidic urine is a major determinant of uric acid urolithiasis).
3. History of gout.
4. History of stroke or myocardial infarction.
5. History of symptomatic coronary artery disease (e.g. angina pectoris) or symptomatic peripheral arterial disease within 1 year prior to Screening.
6. Symptomatic congestive heart failure with a documented ejection fraction below 45%.
7. Poorly controlled arterial hypertension (SBP>160mmHg or DBP>100mmHg at Screening).
8. Women who are pregnant or lactating.
9. The presence of unstable psychiatric disease, cognitive impairment, or dementia that would impair ability of the subject to provide informed consent, according to Site Investigator judgment, or a history of active substance abuse within the prior year.
10. Anything that, in the opinion of the Site Investigator, would place the subject at increased risk or preclude the subject's full compliance with or completion of the study.
11. Use of the following within 30 days prior to Screening: inosine, allopurinol, probenecid, more than 300mg vitamin C daily (note that a subject may take a standard multivitamin up to one tablet or capsule daily). Use of thiazides is permissible as long as the subject is on a stable dose from 1 week prior to Screening.
12. Known hypersensitivity or intolerability to inosine.
13. Renal insufficiency as defined by eGFR < 60 mL/min/1.73m2 at the time of screening.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2020-01-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sabrina Paganoni, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Paganoni S, Zhang M, Quiroz Zarate A, Jaffa M, Yu H, Cudkowicz ME, Wills AM. Uric acid levels predict survival in men with amyotrophic lateral sclerosis. J Neurol. 2012 Sep;259(9):1923-8. doi: 10.1007/s00415-012-6440-7. Epub 2012 Feb 10. PMID 22323210
- [Background] Atassi N, Berry J, Shui A, Zach N, Sherman A, Sinani E, Walker J, Katsovskiy I, Schoenfeld D, Cudkowicz M, Leitner M. The PRO-ACT database: design, initial analyses, and predictive features. Neurology. 2014 Nov 4;83(19):1719-25. doi: 10.1212/WNL.0000000000000951. Epub 2014 Oct 8. PMID 25298304
- [Background] Parkinson Study Group SURE-PD Investigators; Schwarzschild MA, Ascherio A, Beal MF, Cudkowicz ME, Curhan GC, Hare JM, Hooper DC, Kieburtz KD, Macklin EA, Oakes D, Rudolph A, Shoulson I, Tennis MK, Espay AJ, Gartner M, Hung A, Bwala G, Lenehan R, Encarnacion E, Ainslie M, Castillo R, Togasaki D, Barles G, Friedman JH, Niles L, Carter JH, Murray M, Goetz CG, Jaglin J, Ahmed A, Russell DS, Cotto C, Goudreau JL, Russell D, Parashos SA, Ede P, Saint-Hilaire MH, Thomas CA, James R, Stacy MA, Johnson J, Gauger L, Antonelle de Marcaida J, Thurlow S, Isaacson SH, Carvajal L, Rao J, Cook M, Hope-Porche C, McClurg L, Grasso DL, Logan R, Orme C, Ross T, Brocht AF, Constantinescu R, Sharma S, Venuto C, Weber J, Eaton K. Inosine to increase serum and cerebrospinal fluid urate in Parkinson disease: a randomized clinical trial. JAMA Neurol. 2014 Feb;71(2):141-50. doi: 10.1001/jamaneurol.2013.5528. PMID 24366103
- [Derived] Beukenhorst AL, Burke KM, Scheier Z, Miller TM, Paganoni S, Keegan M, Collins E, Connaghan KP, Tay A, Chan J, Berry JD, Onnela JP. Using Smartphones to Reduce Research Burden in a Neurodegenerative Population and Assessing Participant Adherence: A Randomized Clinical Trial and Two Observational Studies. JMIR Mhealth Uhealth. 2022 Feb 4;10(2):e31877. doi: 10.2196/31877. PMID 35119373

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants age 18 and older who met the El Escorial criteria of possible, laboratory-supported probable, probable, or definite criteria for a diagnosis of ALS were recruited across three Northeast ALS Consortium (NEALS) Centers.
Pre-assignment Details: According to the study protocol all participants who consent to the study are considered enrolled. 23 consented participants were deemed ineligible during screening procedures and 2 withdrew consent. Of the 23 ineligible participants, 13 did not meet inclusion criteria and 10 were ineligible due to meeting exclusion criteria.
Period: Overall Study
Arm/Group | Inosine | Placebo
Started | 14 | 9
Completed | 12 | 7
Not Completed | 2 | 2
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Inosine | Placebo | Total
Number analyzed (Participants) | 14 | 9 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 9 | 20
  >=65 years | 3 | 0 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.0 (9.9) | 56.4 (10) | 58.6 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 4 | 14
  Male | 4 | 5 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 13 | 9 | 22
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 14 | 9 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 9 | 23
Amyotrophic Lateral Sclerosis Functional Rating Scale Total Score [Mean (Standard Deviation); unit: units on a scale] — The Amyotrophic Lateral Sclerosis Functional Rating Scale (ALSFRS) is an instrument for evaluating the functional status of patients with Amyotrophic Lateral Sclerosis. It can be used to monitor functional change in a patient over time. It measures across 12 domains with scales in each domain ranging from 0 to 4 with a lower score indicating a more severe deficiency in that domain. The scores across domains are summed to indicate severity of disease as follows: >40 (minimal to mild)
  39-30 (mild to moderate)
  < 30 (moderate to severe)
  < 20 (advanced disease)
  units on a scale | 35.1 (8.4) | 36.6 (6.8) | 35.7 (7.7)
Amyotrophic Lateral Sclerosis Functional Rating Scale Bulbar Subdomain [Mean (Standard Deviation); unit: units on a scale] — The Amyotrophic Lateral Sclerosis Functional Rating Scale (ALSFRS) Bulbar Subdomain is the subdomain of the full Amyotrophic Lateral Sclerosis Functional Rating Scale encompassing questions on speech, salivation, and swallowing. The questions are summed with a lower score indicating a more severe impairment. Maximum score is 12 and minimum score is 0.
  units on a scale | 8.6 (2.8) | 9.0 (3.2) | 8.8 (2.9)
Amyotrophic Lateral Sclerosis Functional Rating Scale Fine-Motor Subdomain [Mean (Standard Deviation); unit: units on a scale] — The Amyotrophic Lateral Sclerosis Functional Rating Scale (ALSFRS) Fine Motor Subdomain is the subdomain of the full Amyotrophic Lateral Sclerosis Functional Rating Scale encompassing questions on handwriting, cutting food, and dressing and hygiene. The questions are summed with a lower score indicating a more severe impairment. Maximum score is 12 and minimum score is 0.
  units on a scale | 8.5 (3.3) | 8.4 (3.1) | 8.5 (3.1)
Amyotrophic Lateral Sclerosis Functional Rating Scale Gross-Motor Subdomain [Mean (Standard Deviation); unit: units on a scale] — The Amyotrophic Lateral Sclerosis Functional Rating Scale (ALSFRS) Gross Motor Subdomain is the subdomain of the full Amyotrophic Lateral Sclerosis Functional Rating Scale encompassing questions on turning in bed, walking, and climbing stairs. The questions are summed with a lower score indicating a more severe impairment. Maximum score is 12 and minimum score is 0.
  units on a scale | 7.4 (2.7) | 7.7 (2.6) | 7.5 (2.6)
Amyotrophic Lateral Sclerosis Functional Rating Scale Respiratory Subdomain [Median (Standard Deviation); unit: units on a scale] — The Amyotrophic Lateral Sclerosis Functional Rating Scale (ALSFRS) Respiratory Subdomain is the subdomain of the full Amyotrophic Lateral Sclerosis Functional Rating Scale encompassing questions on dyspnea, orthopnea, and respiratory insufficiency. The questions are summed with a lower score indicating a more severe impairment. The maximum score is 12 and minimum score is 0.
  units on a scale | 10.5 (2.5) | 11.4 (0.88) | 10.9 (2.05)
Vital Capacity Percent Predicted Max [Mean (Standard Deviation); unit: percentage predicted] — To measure Vital Capacity, the patient inhales maximally, then exhales as rapidly and as completely as possible. Normal lungs generally can empty more than 80 percent of their volume in six seconds or less. Normal range is 80%-120%. A lower score is indicative of reduced lung capacity.
  percentage predicted | 81.9 (21.8) | 86.1 (29.5) | 83.5 (24.3)
Years from Symptom onset to Screening [Mean (Standard Deviation); unit: years] | 1.97 (1.15) | 2.56 (1.51) | 2.2 (1.3)
Years from Diagnosis to Screening [Median (Standard Deviation); unit: years] | 0.79 (0.73) | 1.47 (1.33) | 1.06 (1.04)
Years from Symptom onset to Diagnosis [Mean (Standard Deviation); unit: years] | 1.18 (1.12) | 1.08 (0.54) | 1.14 (0.92)
Weight [Mean (Standard Deviation); unit: kilograms] | 72.7 (10.3) | 69.7 (17.9) | 71.5 (13.6)
Urate [Mean (Standard Deviation); unit: milligrams per deciliter] | 3.94 (1.11) | 3.96 (0.48) | 3.94 (0.90)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Safety will be assessed by the occurrence of adverse events such as kidney stones and gout (expected adverse events) in all participants receiving at least 1 dose of study drug
Time Frame: Baseline to Week 24
Measure: Number; unit: participants
Arm/Group | Inosine | Placebo
Number analyzed (Participants) | 14 | 9
participants | 11 | 7

2. Primary Outcome: Tolerability to Complete the Entire 20 Week Study on Study Drug
Description: Tolerance of study drug will be defined as the number of participants who able to complete the 20-week study without permanently discontinuing study drug or suspending study drug for greater than 28 days
Time Frame: Baseline to Week 20
Measure: Count of Participants; unit: Participants
Arm/Group | Inosine | Placebo
Number analyzed (Participants) | 14 | 9
Participants | 12 | 7

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the time of first participant consent through final participant's completion of the study. This covered an active study period of 2 years and 3 months. Participants were followed from time of consent through completion of their study participation or withdrawal of consent. Adverse event data was collected for 24 weeks.
Description: Adverse Events classified by MedDRA system organ class, higher level term, and preferred term
Arm/Group | Inosine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/14 | 1/9
Serious Adverse Events (participants affected / at risk) | 4/14 | 1/9
Other Adverse Events (participants affected / at risk) | 11/14 | 7/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inosine (N=14) | Placebo (N=9)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Device Related Infection (Infections and infestations) | 1 (1) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inosine (N=14) | Placebo (N=9)
Anaemia Macrocytic (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Normochromic Normocytic Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Cardiogenic Shock (Cardiac disorders) | 0 (0) | 1 (1)
Eye Pruritus (Eye disorders) | 1 (1) | 0 (0)
Lacrimation Increased (Eye disorders) | 1 (1) | 0 (0)
Abdominal Discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypoaesthesia Oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Implant Site Pain (General disorders) | 1 (1) | 0 (0)
Subcutaneous Abscess (Infections and infestations) | 0 (0) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Eye Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 4 (6) | 0 (0)
Skin Abrasion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Blood Potassium Decreased (Investigations) | 1 (1) | 0 (0)
Electrocardiogram St Segment Elevation (Investigations) | 0 (0) | 1 (1)
Ph Urine Abnormal (Investigations) | 1 (1) | 0 (0)
Platelet Count Decreased (Investigations) | 0 (0) | 1 (2)
Weight Decreased (Investigations) | 0 (0) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dupuytren's Contracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 1 (2)
Muscle Contractions Involuntary (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory Acidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Central Venous Catheterisation (Surgical and medical procedures) | 0 (0) | 1 (1)
Medical Device Removal (Surgical and medical procedures) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-07-01): https://cdn.clinicaltrials.gov/large-docs/11/NCT03168711/Prot_SAP_000.pdf
  • Informed Consent Form (2019-07-01): https://cdn.clinicaltrials.gov/large-docs/11/NCT03168711/ICF_001.pdf